CLINICAL TRIAL: NCT04168138
Title: D-CTAG in the Treatment of Newly Diagnosed Acute Myeloid Leukemia in Elderly Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huihan Wang (Other)
Responsible Party: Sponsor-Investigator, Huihan Wang, Deputy Chief Physician, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HhWang
Record Dates: First submitted 2019-11-10; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: D-CTAG; Acute Myeloid Leukemia; rhTPO
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine; Aclarubicin; Granulocyte Colony-Stimulating Factor; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Newly diagnosed AML in elderly patient (Experimental): D: Decitabine(15mg/m2) d1-5 G: G-CSF（300ug/d） d0-9(stop using when WBC>20*109/L) T: rhTPO(15000U/d) d3,5,7,9, d11- (Platelet>50*109/L) A: Aclarubicin(10mg/d) d3-6 C: Cytarabine(15mg Q12h) d3-9
  Interventions: Drug: rhTPO

INTERVENTIONS:
Drug: rhTPO — D: Decitabine(15mg/m2) d1-5 G: G-CSF（300ug/d） d0-9(stop using when White Blood Cell (WBC)>20*109/L) T: rhTPO(15000U/d) d3,5,7,9, d11- (Platelet>50*109/L) A: Aclarubicin(10mg/d) d3-6 C: Cytarabine(15mg Q12h) d3-9
  Other Names: Decitabine; Aclarubicin; G-CSF; Cytarabine

SUMMARY:
With the aging of society, the incidence of elderly leukemia in China has been increasing year by year. The elderly patients with Acute Leukemia have poor basal state, and there are many important organ diseases such as heart, liver and kidney. The incidence of infection and hemorrhage is high in elderly patients after chemotherapy. These characteristics make the treatment of elderly leukemia difficult. So we propose a new treatment plan by using the therapy that rhTPO may promote the leukemia cells into the division cycle.We use the synergistic effect of G-CSF and rhTPO to promote leukemia cells into the division cycle, thereby the cells can be killed by cytotoxic drugs. At the same time, G-CSF and rhTPO are used to promote the growth of granulocytes and platelets, therefore the side effects of treatment of elderly leukemia can be alleviated. We provide a safe and effective chemotherapy for elderly leukemia patients, so that more elderly patients receive chemotherapy,which has important practical significance.

DETAILED DESCRIPTION:
In China，the incidence of leukemia is 2.76/100,000. Leukemia ranks first in the mortality rate of malignant tumors in children and adults under 35 years old. With the aging of society, the incidence of elderly leukemia in China has been increasing year by year. The elderly patients with Acute Leukemia have poor basal state, and there are many important organ diseases such as heart, liver and kidney. The incidence of infection and hemorrhage is high in elderly patients after chemotherapy. These characteristics make the treatment of elderly leukemia difficult.In 1995, Japanese scholar Yamada proposed the CAG protocol (granulocyte colony-stimulating factor (G-CSF) combined with low-dose cytarabine (Ara-C) and aclacinomycin (ACR)) for the treatment of Acute Myeloid leukemia in elderly patients.when a better response rate was obtained, the side effects were significantly reduced. Although the application of G-CSF in the CAG protocol reduces the incidence of granulocytopenic co-infection in elderly patients, thrombocytopenia, another common side effect of chemotherapy in elderly patients, still limits the efficacy and safety of treatment in elderly patients. Recombinant human thrombopoietin (rhTPO) is approved for thrombocytopenia after solid tumor chemotherapy, but there are few studies on Acute Myeloid Leukemia (AML).So we propose a new treatment plan by using the therapy that rhTPO may promote the leukemia cells into the division cycle.We use the synergistic effect of G-CSF and rhTPO to promote leukemia cells into the division cycle, thereby the cells can be killed by cytotoxic drugs. At the same time, G-CSF and rhTPO are used to promote the growth of granulocytes and platelets, therefore the side effects of treatment of elderly leukemia can be alleviated.Recent studies have found that erythropoietin and G-CSF act on the cardiovascular system.By mobilizing bone marrow stem cells to repair ischemic myocardium,they promote cardiomyocyte regeneration and neovascularization in the ischemic area. In addition to promoting platelet growth, rhTPO can also reduce the cardiotoxicity of anthracyclines in elderly patients with CAG.We provide a safe and effective chemotherapy for elderly leukemia patients, so that more elderly patients receive chemotherapy,which has important practical significance.

The cycle of this trial is 8 cycles.After all the treatments completing, the patients are followed up to observe the bone marrow.In the first year,the patients will be reviewed every 3 months;In the second year ,They will be reviewed every 6 months, and two year later,they will be reviewed every year, including morphological analysis of bone marrow.After the trial is completed, the survival information of the patients will be followed up by telephone or through the trial center every 3 months.

About combined medication:1) During the whole test period, patients are not allowed to receive other anti-tumor measures other than test drugs, including radiotherapy, chemotherapy, targeted therapy, immunological preparation, hematopoietic stem cell transplantation, etc.;2) The investigator can take appropriate supportive treatment after evaluating the relationship between adverse events and trial medication. The start and duration of supportive treatment are recorded in the original record. These treatments include antiemetics, antidiarrheal, antipyretic, antiallergic, diabetes treatment, use of antihypertensive drugs, use of analgesics, use of antibiotics, and other uses such as blood products;3)The patients can be given symptomatic treatment when hematological toxicity is in level 3 or after the investigator has judged the condition, and record in the combined medication;4)The patients can be given symptomatic treatment when non-hematological toxicity is in level 2 and record in the combined medication;5) Basic diseases should be given to maintain treatment;6) All concomitant medications, generic names, medication purposes, dosages, and medication time received by the patient should be fully recorded in the original record;7) It is forbidden to use other clinical trial drugs during the trial.

The use of TPO in new technologies may increase the incidence of thrombosis. In this trial, rhTPO will be discontinued when platelets > 50*109/L. Because of chemotherapy, bone marrow suppression and thrombocytopenia are observed. At the same time, newly diagnosed leukemia often combined with thrombocytopenia. No special medication will be needed to prevent thrombosis, and platelet level should be closely observed. Other technologies, other risks and response plans are the same as traditional treatment plans The cost of patient medication in this trial is similar to that of traditional treatment . The chemotherapy drugs used are all listed drugs

ELIGIBILITY:
Inclusion Criteria:

1. Age 60 or above, male or female;
2. Acute Myeloid Leukemia (non-M3) diagnosed according to the 2008 World Health Organization (WHO) diagnostic criteria for myeloid malignancies;
3. Newly diagnosed, no treatment for anti-leukemia;
4. The Eastern Cooperative Oncology Group（ECOG） status score is 0 to 3 points;
5. Expected survival time ≥ 3 months;
6. No serious heart, lung, liver or kidney disease;
7. History of no thromboembolism
8. Ability to understand and be willing to sign the informed consent form of this trial.

Exclusion Criteria:

1. used to be allergic to the drugs contained in the protocol or to drugs similar in chemical structure to the test drugs;
2. serious active infections;
3. Patients with extramedullary lesions;
4. Patients who use drugs and long-term alcohol abuse to influence the evaluation of test results;
5. Inability to obtain informed consent and cannot complete the trial treatment and examination procedures because of mental illness or other conditions
6. Patients with clinically significant corrected QT interval (QTc) prolongation (male > 450ms, female > 470ms), Ventricular Tachycardia (VT), Atrial Fibrillation (AF), grade II or higher heart block, Myocardial Infarction (MI) within 1 year, Congestive Heart Failure (CHF), coronary heart disease with symptoms who need medical treatment;
7. Abnormal liver function (total bilirubin > 1.5 times the upper limit of normal value, Alanine aminotransferase(ALT) / Aspartate aminotransferase (AST) >2.5 times the upper limit of normal value or ALT / AST in patients with liver invasion > 5 times the upper limit of normal value of normal), abnormal renal function (serum Creatinine > 1.5 times the upper limit of normal);
8. The investigator determine that the participants are not suitable

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival（PFS） | 2 years after the end of treatment of the last patient enrolled
  Progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Huihan Wang, Doctor, Principal Investigator — Shengjing Hospital
Locations (1):
- ShengJing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No